CLINICAL TRIAL: NCT02026219
Title: Comparison of Clopidogrel and Ticagrelor on Microvascular Dysfunction in Acute Coronary Syndrome Patients: The Index of MIcrocirculatory Resistance After PCI in STEMI Patients (TIME Study)
Brief Title: Comparison of Clopidogrel and Ticagrelor on Microvascular Dysfunction in ST-Segment Elevation Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUH-IRB-13-2256
Record Dates: First submitted 2013-12-24; First posted 2014-01-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Non-ST Segment Elevation Myocardial Infarction; ST Segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Experimental): Clopidogrel 600mg loading
  Interventions: Drug: Clopidogrel
- Ticagrelor (Experimental): Ticagrelor 180mg loading
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 600mg loading
  Arms: Clopidogrel
Drug: Ticagrelor — Ticagrelor 180mg loading
  Arms: Ticagrelor

SUMMARY:
Ticagrelor is a non-thienophyridine, direct P2Y12 blocker that is more potent than clopidogrel and is associated with less interindividual variability. In the PLATO trial, it was found to be superior to clopidogrel with respect to cardiovascular outcomes and total mortality without increasing the risk of bleedings.

More potent and reversible receptor bindings are possible explanation for the superior outcomes. Beside the potent effect on inhibition of antiplatelet function, ticagrelor has previously been demonstrated to increase adenosine levels by inhibiting adenosine re-uptake in tissue level and can induce adenosine triphosphate (ATP) release from human red cells, which both stimulate vasodilation of in red blood cells.

ELIGIBILITY:
* Inclusion Criteria:

  * Males and Females
  * between the ages of 18 and 75 years
  * STEMI patients treated with percutaneous coronary intervention
  * Able to provide informed consent
* Exclusion Criteria:

  * History of stroke or transient ischemic attack
  * Platelet count < 100 000/μL
  * Known Bleeding Diathesis
  * Hematocrit <30% or >52%
  * Severe Liver Dysfunction
  * Renal Insufficiency (Creatinine Clearance < 30ml/min)
  * Pregnant females
  * Cardiogenic shock or symptomatic hypotension or sitting SBP < 95 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Index of microcirculatory resistance (IMR) measured after successful coronary intervention | IMR will be immediately assessed after successful PCI patients within 48hr from admission

SECONDARY OUTCOMES:
wall motion score index on three month later TTE from index PCI | TTE will be assessed in all enrolled patients 3 month later from index PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, Incheon, South Korea

REFERENCES:
- [Derived] Park SD, Baek YS, Woo SI, Kim SH, Shin SH, Kim DH, Kwan J, Park KS. Comparing the effect of clopidogrel versus ticagrelor on coronary microvascular dysfunction in acute coronary syndrome patients (TIME trial): study protocol for a randomized controlled trial. Trials. 2014 May 1;15:151. doi: 10.1186/1745-6215-15-151. PMID 24885437